CLINICAL TRIAL: NCT05232461
Title: A Pilot, Open-Label, Randomized, Single-Dose, Three-Treatment, Three-Period Crossover Study to Evaluate the Effect of Food on the Bioavailability of PrimeC-ER Tablets and the Comparative Bioavailability of PrimeC-ER and Ciprofloxacin Tablets and Celecoxib Capsules, When Co-Administered, in Healthy Adult Subjects
Brief Title: A Pilot Study to Evaluate the PK Profile of PrimeC-ER Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroSense Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NST-PK-001
Record Dates: First submitted 2022-01-19; First posted 2022-02-09 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ciprofloxacin; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PrimeC ER Fasted (Active Comparator): Single dose PrimeC-ER (748 mg), administered following an overnight fast of at least 10 hours.
  Interventions: Drug: PrimeC-ER 748 mg
- PrimeC ER Meal (Active Comparator): Single dose PrimeC-ER (748 mg), administered at 30 minutes after the start of a standardized high-fat, high-calorie breakfast that was preceded by an overnight fast of at least 10 hours.
  Interventions: Drug: PrimeC-ER 748 mg
- Marketed ciprofloxacin and celecoxib (Active Comparator): Single dose of 750 mg of ciprofloxacin 200 mg of celecoxib, co-administered following an overnight fast of at least 10 hours.
  Interventions: Drug: Ciprofloxacin 750 MG; Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: PrimeC-ER 748 mg — PrimeC-ER is an extended release formulation of a fixed dose combination of ciprofloxacin and celecoxib
  Arms: PrimeC ER Fasted; PrimeC ER Meal
Drug: Ciprofloxacin 750 MG — Ciprofloxacin
  Arms: Marketed ciprofloxacin and celecoxib
Drug: Celecoxib 200mg — Celecoxib
  Arms: Marketed ciprofloxacin and celecoxib

SUMMARY:
This is an open-label, randomized, single-dose, three treatment, three-period crossover study comparing the test and reference products under fasted or fed conditions (as applicable). In one period of the study, PrimeC-ER tablets will be administered to subjects following an overnight fast of at least 10 hours. In a second period of the study, PrimeC-ER tablets will be administered to subjects at 30 minutes following the start of a standardized high-fat, high-calorie breakfast that was preceded by an overnight fast of at least 10 hours. In a third period of the study, a single 750 mg dose of ciprofloxacin and a single 200 mg dose of celecoxib will be co-administered to subjects following an overnight fast of at least 10 hours. The order of administration will follow a six-sequence randomization schedule. Blood samples will be collected at pre-dose and at intervals over 48 hours after dosing in each study period. Subjects will be confined at the clinical facility from at least 10.5 hours before dosing until 48 hours after dosing in each study period. The interval between doses will be at least 7 days. Subjects will return to the clinical facility 7 days (± 1 day) after the last study drug administration for an end-of study follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-55 years of age, inclusive, with a Body Mass Index (BMI) of 18.5 29.9 kg/m², inclusive.
2. Female subjects must meet at least one of the following criterion:

   * Agree to abstain from sexual intercourse from screening and throughout the duration of the study.
   * Have used and agree to continue to use a reliable method of contraception (e.g., hormonal contraceptives, condom with spermicide, IUD) for at least 30 days before initial dosing and throughout the duration of the study.
   * Surgically sterile (bilateral oophorectomy or hysterectomy, bilateral tubal ligation at least 3 months before initial dosing or Essure® device placement before the year 2018).
   * At least 1 year postmenopausal and have a documented FSH level ≥ 40 mIU/mL at screening.
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations.
5. Subject understands the requirements of the study and is willing to comply with all study requirements.

Exclusion Criteria:

1. Females who are pregnant, lactating or likely to become pregnant during the study.
2. History of allergy or hypersensitivity to ciprofloxacin or other fluoroquinolones, celecoxib or other NSAIDs, any component of the study products, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction especially cardiovascular disorders (e.g., hearth failure, edema), respiratory disorders (e.g., asthma), hypertension, renal or hepatic disorders, diabetes or obesity.
4. QTc interval > 450 msec for males or > 470 msec for females or any clinically significant ECG abnormalities that, in the Investigator's opinion, would compromise the subject's safety for inclusion in the study. Significant history or current evidence of risk factors for Torsade de Pointes (TdP) (e.g., cardiac disease, heart failure, clinically significant hypokalemia or other electrolyte disorders, family history of Long QT Syndrome), as determined by the Investigator.
5. History or current evidence of myasthenia gravis or myasthenic syndrome.
6. History or current evidence of epilepsy, other seizures disorders, or other risk factors that may predispose to seizures or lower the seizure threshold; tendinitis or tendon rupture; peripheral neuropathy or aortic aneurysms.
7. Significant acute illness (e.g. acute infection) within 14 days before initial dosing, as determined by the Investigator.
8. Clinically significant history or presence of gastrointestinal disease (e.g., peptic ulcer, gastrointestinal bleeding) or history of malabsorption within the last year, as determined by the Investigator.
9. History of psychiatric disorders (e.g., anxiety, depression, insomnia, confusion) occurring within the last two years, which required the subject to be hospitalized or treated with medication.
10. Presence of a medical condition requiring regular treatment with prescription drugs (except hormonal contraceptives).
11. Use of pharmacologic agents (prescription or over-the-counter) or herbal products known or suspected to induce or inhibit drug-metabolizing enzymes (especially inducers and inhibitors of CYP1A2 and CYP2C9) within 30 days before initial dosing.
12. Use of dietary products (e.g., grapefruit products of all types) known or suspected to induce or inhibit drug-metabolizing enzymes (especially inducers and inhibitors of CYP1A2 and CYP2C9) within 14 days before initial dosing.
13. Use of any prescription medications (other than hormonal contraceptives and those noted above), especially prescription medications implicated in TdP or cardiac arrhythmia, terfenadine, pimozide, ergotamine; dihydroergotamine or over-the-counter medications implicated in TdP or cardiac arrhythmia; medications that interfere with hemostasis (e.g., warfarin, selective serotonin reuptake inhibitors, selective serotonin norepinephrine reuptake inhibitors), other quinolones, digoxin, and NSAIDs or antibiotics (all dosage forms and routes of administration; other than the study drugs) within 14 days before initial dosing.
14. Known or suspected to be a poor CYP2C9 metabolizer.
15. Receipt of any drug as part of a research study within 30 days before initial dosing or 5 half-lives, whichever is longer.
16. Drug or alcohol addiction, as determined by the Investigator, in the 12 months before initial dosing.
17. History of excessive alcohol consumption (on average more than 14 units of alcohol/week) during the past 12 months.
18. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days before initial dosing.
19. Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
20. Positive test results for drugs of abuse at screening.
21. If female, has a positive pregnancy test at screening.
22. Use of tobacco- or nicotine-containing products within 90 days before initial dosing.
23. Difficulty swallowing capsules or tablets whole.
24. Unable or unwilling to comply with protocol restrictions and required study procedures (including consuming the entire high-fat, high-calorie breakfast).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | 1 month
  AUC is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
AUC 0-∞ | 1 month
  AUC is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
Cmax | 1 month
  Cmax is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.

SECONDARY OUTCOMES:
Tmax | 1 month
  Tmax is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
Tlag | 1 month
  Tlag is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
λz | 1 month
  λz is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
T1/2 | 1 month
  T1/2 is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
R^2 | 1 month
  R^2 is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.
AUC %extrap | 1 month
  AUC %extrap is tested in order to assess the effect of food on the bioavailability of PrimeC-ER Tablets (748 mg) in healthy adult male and female subjects, and in order to evaluate the comparative bioavailability of PrimeC-ER Tablets (748 mg) relative to a 750 mg dose of ciprofloxacin tablets and a 200 mg dose of celecoxib capsules, when co-administered, under fasted conditions in healthy adult male and female subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Novum, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No